CLINICAL TRIAL: NCT06694922
Title: Turkish Validity and Reliability Study of the Adult Food and Nutrition Literacy Assessment Tool
Brief Title: Turkish Validation of the Adult Nutrition Literacy Tool
Status: Completed | Type: Observational
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Principal Investigator, Emine Elibol, Assist. Prof., Ankara Yildirim Beyazıt University
Other Study IDs: AYBUELİBOL005
Record Dates: First submitted 2024-11-09; First posted 2024-11-19 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-10

CONDITIONS: Nutrition
Keywords: Validity and Reliability; Nutrition; Food

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Young people: This study evaluated the validity and reliability of the Food and Nutrition Literacy Assessment Tool (FNLAT) in a sample of 849 Turkish adults. Reliability was tested using Cronbach's alpha, test-retest, and Pearson correlation, while construct validity was analyzed via factor analysis. Data were processed with SPSS and AMOS software.

SUMMARY:
This study evaluated the validity and reliability of the Food and Nutrition Literacy Assessment Tool (FNLAT) in a sample of 849 Turkish adults. Reliability was tested using Cronbach's alpha, test-retest, and Pearson correlation, while construct validity was analyzed via factor analysis. Data were processed with SPSS and AMOS software.

DETAILED DESCRIPTION:
Aim: The aim of this study is to evaluate the validity and reliability of the Food and Nutrition Literacy Assessment Tool in Turkey.

Subject and Methods: The study included 849 individuals aged 19-64 years (316 males, 563 females). A questionnaire containing socio-demographic characteristics and the " Food and Nutrition Literacy Assessment Tool (FNLAT)" and " General Nutrition Knowledge Questionnaire (GNKQ)" were used as data collection tools. Test-retest was performed on 60 individuals at 3-week intervals. Cronbach's alpha, test-retest, and Pearson correlation analyses were conducted to assess the reliability of the scale. The construct validity of the scale was determined using explanatory factor analysis. The data were analyzed using the SPSS (Statistical Package for Social Sciences) for Windows 25.0 and AMOS 21 programs.

ELIGIBILITY:
Inclusion Criteria:

* People aged 19 to 64 years

Exclusion Criteria:

* Individuals diagnosed with psychiatric or neurological diseases
* Individuals with alcohol or drug addiction.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community sample in Ankara and Elazığ, Turkey
Sampling Method: Probability Sample
Enrollment: 849 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
General Nutrition Knowledge Questionnaire (GNKQ) Assessment | Basaline
  The General Nutrition Knowledge Questionnaire was developed to measure general nutrition knowledge, with Turkish validity and reliability established. This questionnaire consists of 35 questions in four sub-components: nutrition recommendations (11 questions), nutrition knowledge (70 questions), food selection (11 questions), and diet-disease relationship (35 questions). Each correct answer within these sub-components is scored as '1,' while incorrect and unsure responses are scored as '0.' The total score ranges from a minimum of 0 to a maximum of 127, with higher scores indicating a greater level of nutrition knowledge. Permission was obtained from the authors
Food and Nutrition Literacy Assessment Tool (FNLAT) Assessment | Basaline
  The Food and Nutrition Literacy Assessment Tool was designed to measure food and nutrition literacy, with an internal validity index of ≥90% confirming its content validity. The tool includes six factors: one in the knowledge domain (nutrition knowledge) and five in the skills domain (functional skills, interactive skills, advocacy, critical information analysis, and food label reading skills). Confirmatory factor analysis indicated acceptable model fit indices, validating the construct of FNLAT. Cronbach's Alpha and intraclass correlation coefficient (ICC) values confirmed the internal consistency and stability over time. Scoring: FNLAT scores are calculated by summing raw scores for each subscale or the total, then converting them to a 0-100 scale, where higher scores indicate greater food and nutrition literacy.

SECONDARY OUTCOMES:
Sociodemographic characteristics | Basaline
  Sociodemographic characteristics will be assessed using a structured questionnaire developed by the researchers. The questionnaire will include items measuring age, gender, education level, and income status. The results will be presented as numbers and percentages for each characteristic
Body Mass Index (BMI) | Basaline
  Kilograms per square meter (kg/m2)
Body weight | Basaline
  Body weight in kg
Height | Basaline
  Height in cm

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Yıldırım Beyazıt University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No